CLINICAL TRIAL: NCT02179021
Title: Is Haemostasis Impaired in Cardiac Arrest Patients During Therapeutic Hypothermia?
Brief Title: Haemostasis and Therapeutic Hypothermia
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-0022
Record Dates: First submitted 2014-06-12; First posted 2014-07-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2014-06

CONDITIONS: Hypothermia; Heart Arrest
Keywords: Thromboelastometry; Haemostasis; Hypothermia; Heart arrest
MeSH Terms: conditions — Hypothermia; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate, if the haemostasis is impaired in cardiac arrest patients during therapeutic hypothermia compared with normothermia.

DETAILED DESCRIPTION:
Treatment with mild therapeutic hypothermia, 32-34 °C for 12-24 hours, has shown to improve the neurologic outcome in comatose survivors of out-of-hospital cardiac arrest. Hypothermia is suspected to inhibit haemostasis and therefore cardiac arrest patients with a risk of bleeding are not treated with therapeutic hypothermia. However, the impact on the coagulation system during mild therapeutic hypothermia, has not yet been fully investigated.

The investigators aim to investigate if mild therapeutic hypothermia influences haemostasis. We are including survivors of cardiac arrest, who are treated with hypothermia for 24-48 hours.

Blood will be sampled during hypothermia and secondly during normothermia. 30 minutes after the blood are sampled it will be analyzed using a sensitive low-tissue-factor assay with rotational thromboelastometry (ROTEM®). All the dynamic coagulation parameters obtained on the ROTEM® at hypothermia and normothermia, respectively, will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with therapeutic hypothermia, for minimum 24 and up to 48 hours, due to cardiac arrest.

Exclusion Criteria:

* age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with mild therapeutic hypothermia for 24-48 hours due to cardiac arrest.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To detect changes in clotting time in seconds (s), during the first 3 days after target temperature (34 °C) is reached. | 22, 46 and 70 hours after target temperature (34 °C) is reached (+/- 2 hours).
  Clotting time will be measured by thromboelastometry on the ROTEM-analyzer using a low-tissue-factor assay.

SECONDARY OUTCOMES:
To detect changes in the clot formation time (s), during the first 3 days after target temperature (34 °C) is reached. | 22, 46 and 70 hours after target temperature (34 °C) is reached (+/- 2 hours).
  Coagulation parameters will be measured by thromboelastometry on the ROTEM® using a low-tissue-factor assay.
To detect changes in maximum clot firmness (mm), during the first 3 days after target temperature (34 °C) is reached. | 22, 46 and 70 hours after hypothermia is reached. (+/- 2 hours)
  Coagulation parameters will be measured by thromboelastometry on the ROTEM® using a low-tissue-factor assay.
To detect changes in time to maximum velocity (s), during the first 3 days after target temperature (34 °C) is reached. | 22, 46 and 70 hours after target temperature (34 °C) is reached (+/- 2 hours).
  Coagulation parameters will be measured by thromboelastometry on the ROTEM® using a low-tissue-factor assay.
To detect changes in maximum velocity (mm/min.), during the first 3 days after target temperature (34 °C) is reached. | 22, 46 and 70 hours after target temperature (34 °C) is reached (+/- 2 hours).
  Coagulation parameters will be measured by thromboelastometry on the ROTEM® using a low-tissue-factor assay.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, PhD, Study Director — University of Aarhus; Anne Katrine Wulff Nielsen, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Department of Clinical Biochemistry and Dept of Anethesiology and Intensive Care., Aarhus N, Denmark

REFERENCES:
- [Derived] Nielsen AK, Jeppesen AN, Kirkegaard H, Hvas AM. Changes in coagulation during therapeutic hypothermia in cardiac arrest patients. Resuscitation. 2016 Jan;98:85-90. doi: 10.1016/j.resuscitation.2015.11.007. Epub 2015 Nov 22. PMID 26593973